CLINICAL TRIAL: NCT06818734
Title: Implementation of a Clinical Decision Support Tool for Postpartum Depression
Acronym: CDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-03027259
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Postpartum Depression
Keywords: Clinical decision support tool
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention: CDS support , clinician (Experimental): Clinicians in the intervention arm will refer patients based on the CDS.The CDS will alert clinicians only if patients have high risk of developing PPD, and provide clinicians with risk score, risk factors, and anticipatory actions with an order set to assist with ordering. Clinicians will make the ultimate clinical judgement after receiving CDS aid, including taking no actions towards PPD prevention. Clinicians will manage patients per usual care, including initiating PPD preventive such as conducting referrals to nutrition and behavioral health, suggest educational readings through patient portals, or no actions.
  Interventions: Other: Clinical Decision Support Tool
- No intervention: Patients (No Intervention): The CDS will alert clinicians only if patients have high risk of developing PPD. Clinicians will manage patients per usual care, including initiating PPD preventive such as conducting referrals to nutrition and behavioral health, suggest educational readings through patient portals, or no actions.
- Intervention: Patients (Experimental)
  Interventions: Other: Clinical Decision Support Tool

INTERVENTIONS:
Other: Clinical Decision Support Tool — The CDS in and AI algorithm that will alert clinicians only if patients have high risk of developing PPD, and provide clinicians with risk score, risk factors, and anticipatory actions with an order set to assist with ordering. Clinicians will make the ultimate clinical judgement after receiving CDS aid, including taking no actions towards PPD prevention. Clinicians will manage patients per usual care, including initiating PPD prevention such as conducting referrals to nutrition and behavioral health, suggest educational readings through patient portals, or no actions. Clinicians in the intervention arm will refer patients based on the CDS.
  Arms: Intervention: CDS support , clinician; Intervention: Patients

SUMMARY:
This study will evaluate the use of an automated process in the electronic health record (EHR) that will help providers to detect patients at risk of developing postpartum depression (PPD).

DETAILED DESCRIPTION:
The goal of this randomized clinical trial is to assess the implementation of a clinical decision support (CDS) tool. The tool is designed to assist providers in managing patients at risk of developing of postpartum depression.

Investigators hypothesize that this tool will be acceptable and feasible for use and improve the use of mental health services for postpartum depression.

Patients in the control arm will receive usual care, while those in the intervention arm will receive CDS.

Clinicians will manage patients per usual care, including initiating PPD preventive such as conducting referrals to nutrition and behavioral health, suggest educational readings through patient portals, or no actions. Clinicians in the intervention arm will refer patients based on the CDS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* being seen at one of participating clinics
* pregnancy at 20 week gestation or more

Exclusion Criteria:

* Does not speak inclusion
* does not have internet access

Clinician eligibility:

* If they manage patients in the three clinics as a board-certified OBGYN clinician.
* No exclusion criteria apply for clinician based on their knowledge and experience in treating PPD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability as measured by Unified Theory of Technology Acceptance Theory (UTAUT). | One month after initiation of tool use and three months after use.
  UTAUT has five constructs: performance expectation, effort expectation, social influence, facilitating conditions, and behavioral intention. The performance expectation construct in UTAUT is the CDS's ability to identify patients at risk of PPD that clinicians agree with. For each construct, responses will be sought in the 7-point Likert scale, setting 1 as 'strongly disagree', 2 as 'disagree', to 7 as 'strongly agree'. We will average the acceptability survey responses at the end of the study for each of the 5 UTAUT constructs to create a binary variable. An average score of 5 or above will be considered acceptance and non-acceptance otherwise
Appropriateness as measured by Appropriateness Measure (IAM). | One month after initiation of tool use and three months after use.
  IAM is a 4-item measure to assess the appropriateness of the intervention, respectively, with excellent usability. IAM is to be answered by participants in 5-point response scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree.
Feasibility as measured by Feasibility of Intervention Measure (FIM). | One month after initiation of tool use and three months after use.
  FIM is a 4-item measure to assess the feasibility of the intervention, respectively, with excellent usability. FIM is to be answered by participants in 5-point response scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree.
Mental Health service utilization as measured by number of mental health visits | one month and three month
  Mental health service utilization includes presentations to ED or inpatient admission for mental health related reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Yiye Zhang, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Center for Community Health: 515 6th street (3rd floor), Brooklyn, New York
  - Ob GYN Lower Manhattan 156 William street, New York City, New York, New York
  - Weill Cornell Medicine- Women's Health practice 505 East 70th street, New York City, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The study protocol with the statistical analysis plan will be available following publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available once published.
Access Criteria: Anyone who subscribes to the journal, or has access online will be able to review the data.

REFERENCES:
- [Background] Krause N, Borawski-Clark E. Social class differences in social support among older adults. Gerontologist. 1995 Aug;35(4):498-508. doi: 10.1093/geront/35.4.498. PMID 7557520
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Zhang Y, Wang S, Hermann A, Joly R, Pathak J. Development and validation of a machine learning algorithm for predicting the risk of postpartum depression among pregnant women. J Affect Disord. 2021 Jan 15;279:1-8. doi: 10.1016/j.jad.2020.09.113. Epub 2020 Sep 30. PMID 33035748
- [Background] Wang S, Pathak J, Zhang Y. Using Electronic Health Records and Machine Learning to Predict Postpartum Depression. Stud Health Technol Inform. 2019 Aug 21;264:888-892. doi: 10.3233/SHTI190351. PMID 31438052
- [Background] Venkatesh KK, Nadel H, Blewett D, Freeman MP, Kaimal AJ, Riley LE. Implementation of universal screening for depression during pregnancy: feasibility and impact on obstetric care. Am J Obstet Gynecol. 2016 Oct;215(4):517.e1-8. doi: 10.1016/j.ajog.2016.05.024. Epub 2016 May 20. PMID 27210067
- [Background] Dunkel Schetter C, Tanner L. Anxiety, depression and stress in pregnancy: implications for mothers, children, research, and practice. Curr Opin Psychiatry. 2012 Mar;25(2):141-8. doi: 10.1097/YCO.0b013e3283503680. PMID 22262028
- [Background] Cox EQ, Sowa NA, Meltzer-Brody SE, Gaynes BN. The Perinatal Depression Treatment Cascade: Baby Steps Toward Improving Outcomes. J Clin Psychiatry. 2016 Sep;77(9):1189-1200. doi: 10.4088/JCP.15r10174. PMID 27780317
- [Background] Werner E, Miller M, Osborne LM, Kuzava S, Monk C. Preventing postpartum depression: review and recommendations. Arch Womens Ment Health. 2015 Feb;18(1):41-60. doi: 10.1007/s00737-014-0475-y. Epub 2014 Nov 25. PMID 25422150
- [Background] Curtin SC, Abma JC, Ventura SJ, Henshaw SK. Pregnancy rates for U.S. women continue to drop. NCHS Data Brief. 2013 Dec;(136):1-8. PMID 24314113